CLINICAL TRIAL: NCT01771406
Title: Effects of Continuous Positive Airway Pressure (CPAP) and Nebivolol Treatment on Arterial Blood Pressure and Endothelial Function in Hypertensive OSA Patients.
Brief Title: CPAP and Nebivolol in Hypertensive Obstructive Sleep Apnea (OSA) Patients.
Acronym: NEBOSA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: S54613
Record Dates: First submitted 2012-09-05; First posted 2013-01-18 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2012-08

CONDITIONS: Hypertension; Endothelial Dysfunction; Obstructive Sleep Apnea
MeSH Terms: conditions — Hypertension; Sleep Apnea, Obstructive | interventions — Nebivolol; Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nebivolol then CPAP (Experimental): 8 weeks of Nebivolol treatment (5m/day), 6 weeks of washout, 8 weeks of CPAP and if the patient is still hypertensive 8 weeks of Nebivolol plus CPAP treatment
  Interventions: Drug: Nebivolol; Device: Continuous positive airway pressure (CPAP)
- CPAP then Nebivolol (Experimental): 8 weeks of CPAP treatment, 6 weeks of washout, 8 weeks of Nebivolol and if the patient is still hypertensive 8 weeks of Nebivolol plus CPAP treatment
  Interventions: Drug: Nebivolol; Device: Continuous positive airway pressure (CPAP)

INTERVENTIONS:
Drug: Nebivolol — 8 weeks of Nebivolol treatment (5mg/day)
Device: Continuous positive airway pressure (CPAP) — 8 weeks of CPAP treatment
  Other Names: Philips Respironics Remstar System One

SUMMARY:
The aim of this study is to examine how effective CPAP treatment and treatment with nebivolol are respectively on reducing blood pressure and on endothelial dysfunction in patients suffering from obstructive sleep apnea and hypertension.

ELIGIBILITY:
Inclusion Criteria:

* male/female ≥ 18 years old
* patient with obstructive sleep apnea (apnea-hypopnea index ≥ 20) naïve for CPAP treatment
* patient with weak or moderate hypertension (140 <= systolic blood pressure (SBP) < 180 mmHg and 90 <= diastolic blood pressure (DBP) < 110 mmHg naïve for any antihypertensive treatment
* negative pregnancy test
* ambulatory patient
* patient who have signed the informed consent form
* patient affiliated to social security

Exclusion Criteria:

* pregnant or nursing woman
* acute hepatic failure, biliary cirrhosis, cholestasis
* clearance of Cockcroft < 30 ml/min/1.73m2
* sick sinus syndrome, including sino-atrial block
* second and third degree heart block (without a pacemaker)
* history of bronchospasm and bronchial asthma
* bradycardia (heart rate< 60bpm prior to start therapy)
* severe peripheral circulatory disturbances
* acute hypertension (SBP>= 180 mmHg and/or DBP >= 110 mmHg)
* severe daytime sleepiness (Epworth rating scale > 15)
* known cardiovascular pathologies
* contraindication to CPAP
* allergy to nebivolol
* patient treated with antihypertensive drug(s), with class I antiarrhythmics (quinidine, hydroquinidine, cibenzoline, flecainide, disopyramide, lidocaine, mexiletine, propafenone)
* patient treated with CPAP
* patient kept in detention, major protected by the law, hospitalised person
* patient currently participating in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2013-02; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
change in mean arterial blood pressure | measurement assessed at w8,w14,w22

SECONDARY OUTCOMES:
change in endothelial function | measurement assessed at w8,w14,w22

CONTACTS AND LOCATIONS:
Overall Officials: Catharina Belge, M.D., Ph.D., Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Belgium